CLINICAL TRIAL: NCT06589739
Title: Drainage Thoracique Assisté Par Un Casque De Réalité Virtuelle
Brief Title: Chest Drain Insertion Assisted by Virtual Reality
Acronym: CASVIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, STREIT Arthur, Doctor, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A01192-45
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pneumothorax Spontaneous Primary; Pneumothorax Spontaneous Secondary; Pleural Effusion
Keywords: virtual reality; chest drain; pain management; chest tube; anxiety management
MeSH Terms: conditions — Pneumothorax; Pleural Effusion; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality headset (Experimental): Patients in this arm will have a reality helmet placed during chest drain insertion
  Interventions: Device: Virtual Reality Headset
- control group (No Intervention)

INTERVENTIONS:
Device: Virtual Reality Headset — A virtual reality headset will be placed on patients' head before and during chest drain insertion
  Arms: virtual reality headset

SUMMARY:
Clinical study aiming to investigate the potential benefit of the use of virtual reality helmet as a distractor during chest drain insertion to alleviate patients' pain and anxiety

ELIGIBILITY:
Inclusion Criteria:

* Indication of chest drain insertion for pleural effusion or primary spontaneous pneumothorax
* Patient who received clear and loyal information abotu the study protocol
* Patient who consented to participate to the study
* Patient aged 18 years old or older
* Patient affiliated to the french health system

Exclusion Criteria:

* Patient aged less than 18 years old
* Patient in emergency situation
* Patient with severe heart condition
* Patient allergic to silicone
* Patient with severe psychiatric or mental disorder
* patient with binocular vision anomaly
* patient with pacemaker or defibrillator
* patient wearing a hearing aid that cannot be removed
* Patients under the influence of alcohol or drugs, nausea, fatigue, emotional or anxiety disorders, migraine, headaches, infectious disease
* Patient with past medical history of epilepsia or convulsion

  -- Persons covered by articles L. 1121-5 and L1121-8 of the French Public Health Code:
  * Pregnant, parturient or breast-feeding women,
  * Persons of full age subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
  * adults unable to give their consent
  * Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care under articles L. 3212-1 and L. 3213-1.
* Person able to give consent but unable to write
* Person able to give consent but unable to read French
* Patient unable to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain - Chest drain | During chest drain insertion
  Visual Analogic Scale

SECONDARY OUTCOMES:
Pain - Antalgic consumption | during the 24 hours after chest drain insertion
  Antalgic consumption
Pain - 30 minutes | 30 minutes after chest drain insertion
  Visual Analogic scale
Anxiety - Chest drain | During chest drain insertion
  Anxiety Visual Analogic Scale
Anxiety - 30 minutes | 30 minutes after chest drain insertion
  Anxiety Visual Analogic Scale
feasibility | During chest drain insertion
  Was the chest drain insertion duable with the virtual reality headset

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Indovina P, Barone D, Gallo L, Chirico A, De Pietro G, Giordano A. Virtual Reality as a Distraction Intervention to Relieve Pain and Distress During Medical Procedures: A Comprehensive Literature Review. Clin J Pain. 2018 Sep;34(9):858-877. doi: 10.1097/AJP.0000000000000599. PMID 29485536
- [Background] Perenic E, Grember E, Bassard S, Koutlidis N. Impact of virtual reality on pain management in transrectal MRI-guided prostate biopsy. Front Pain Res (Lausanne). 2023 Oct 2;4:1156463. doi: 10.3389/fpain.2023.1156463. eCollection 2023. PMID 37854306